CLINICAL TRIAL: NCT03712488
Title: Differential Expression of CD200 in B-chronic Lymphoproliferative Disorders by Multicolour Flow Cytometry
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Menna-allah M. Atef, Resident doctor, Assiut University
Other Study IDs: flow cytometry in neoplasms
Record Dates: First submitted 2018-10-17; First posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Neoplasms
Keywords: chronic lymphoproliferative disorders
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: flowcytometry — four colour flowcytometry

SUMMARY:
The investigator's goals in this study are to assess :

1. Differential expression of CD200 by using flow cytometric immune-phenotyping in broad range of patients with B-chronic lymphoproliferative disorders (B-CLPD)
2. Role of CD200 in diagnosis , classification and potential value in differential diagnosis
3. CD200 expression level at different anatomic sites

DETAILED DESCRIPTION:
B-Chronic lymphoproliferative disorders (B-CLPDs) are heterogeneous group of disorders with variable clinical presentations and outcomes. They are classified into : chronic lymphocytic leukaemia (CLL), B-cell prolymphocytic leukaemia (B-PLL), hairy cell leukaemia (HCL), and mantle cell lymphoma (MCL), marginal zone lymphoma (MZL), follicular lymphoma (FL) and lymphoplasmacytic lymphoma/WaldenstrÖm macroglobulinaemia (LPL/WM) in leukaemia phase.

Characterization of CLPDs by immunophenotyping (IPT) has become an important and widely used method in hematology. Immunophenotyping is indispensable for the diagnosis of B-CLPDs through recognition of restricted light chain expression and characteristic phenotypes of separate entities.

Immunophenotypic characterization of lymphoid neoplasms is important for diagnosis, sub-classification, and staging and can also play a role in monitoring minimal residual disease. However, the differential diagnosis may be difficult to resolve in some cases, for example, between B-cell neoplasms with full or partial CD5 expression.

CD200 has recently been identified as a potentially useful antigen for flow cytometric immunophenotyping of lymphoid neoplasms, particularly those of the B lineage.

CD200 belongs to the immunoglobulin superfamily and is composed of a light chain-like structure with two extracellular variable- and constant-like domains followed by a transmembrane segment and a cytoplasmic tail.5 CD200 is expressed by various cell types, including B cells, a subset of T cells (including activated T cells), thymocytes, endothelial cells, and neurons .

CD200 generates an immunosuppressive signal by binding to its cognate receptor, CD200 receptor 1 (CD200R1) , which is expressed specifically in granulocytes and monocytes and in a subset of T cells. CD200 appears to play a role in the regulation of antitumor activity and these findings are the basis for ongoing clinical trials using anti-CD200 therapy for chronic lymphocytic leukemia (CLL)

ELIGIBILITY:
Inclusion Criteria:

* All newly diagnosed patients with B-chronic lymphoproliferative disorders

Exclusion Criteria:

* 1) Patient refusal 2) Patients diagnosed T-cell non-hodgkins lymphoma 3) Patients receiving chemo and/or radiotherapy 4) Patients on steroid therapy for any other cause 5) Patients receiving any immunosuppressive drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All newly diagnosed patients with B-chronic lymphoproliferative disorders
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-12-15 (Estimated); Primary Completion 2020-08-30 (Estimated); Study Completion 2021-04-01 (Estimated)

PRIMARY OUTCOMES:
Differential expression of CD200 by using flow cytometric immune-phenotyping in B-chronic lymphoproliferative disorders (B-CLPD) | baseline
  Analysis of expression of CD200 in B-CLPDs for differential diagnosis of subtypes of B-CLPDs

CONTACTS AND LOCATIONS:
Overall Officials: douaa M Sayed, professor, Study Director — South Egypt Cancer Institute

REFERENCES:
- [Background] Ugo V, Leporrier N, Salaun V, Letestu R, Radford-Weiss I, Ramond S, Nataf J, Guesnu M, Picard F, Brouzes C, Perrot JY, Valensi F, Levy V, Ajchenbaum-Cymbalista F, Troussard X. Deciphering leukemic B-cell chronic lymphoproliferative disorders. Leuk Lymphoma. 2006 Oct;47(10):2088-95. doi: 10.1080/10428190600727939. PMID 17071481
- [Background] Schlette E, Fu K, Medeiros LJ. CD23 expression in mantle cell lymphoma: clinicopathologic features of 18 cases. Am J Clin Pathol. 2003 Nov;120(5):760-6. doi: 10.1309/XV4A-G7EM-WQU7-ER67. PMID 14608904
- [Background] Baseggio L, Traverse-Glehen A, Petinataud F, Callet-Bauchu E, Berger F, Ffrench M, Couris CM, Thieblemont C, Morel D, Coiffier B, Salles G, Felman P. CD5 expression identifies a subset of splenic marginal zone lymphomas with higher lymphocytosis: a clinico-pathological, cytogenetic and molecular study of 24 cases. Haematologica. 2010 Apr;95(4):604-12. doi: 10.3324/haematol.2009.011049. Epub 2009 Dec 16. PMID 20015887
- [Background] Challagundla P, Medeiros LJ, Kanagal-Shamanna R, Miranda RN, Jorgensen JL. Differential expression of CD200 in B-cell neoplasms by flow cytometry can assist in diagnosis, subclassification, and bone marrow staging. Am J Clin Pathol. 2014 Dec;142(6):837-44. doi: 10.1309/AJCPBV9ELXC0ECVL. PMID 25389338
- [Background] Rygiel TP, Karnam G, Goverse G, van der Marel AP, Greuter MJ, van Schaarenburg RA, Visser WF, Brenkman AB, Molenaar R, Hoek RM, Mebius RE, Meyaard L. CD200-CD200R signaling suppresses anti-tumor responses independently of CD200 expression on the tumor. Oncogene. 2012 Jun 14;31(24):2979-88. doi: 10.1038/onc.2011.477. Epub 2011 Oct 24. PMID 22020332